CLINICAL TRIAL: NCT04030390
Title: The Influence of Acute Physical Fatigue on Different Balance Tests and Brain Activity During These Balance Tests in a Healthy Population
Brief Title: The Effect of Physical Fatigue on Different Balance Tests and Brain Activity in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Professor Dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 143201939780
Record Dates: First submitted 2019-07-18; First posted 2019-07-24 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Physical Fatigue; Return to Sport; Injury Prevention; EEG; Brain Activity; Balance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Fatigue Condition (Experimental)
  Interventions: Behavioral: Physical Fatigue
- Control Condition (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Physical Fatigue — Maximal cycling effort for 30s (Wingate modified)
  Arms: Physical Fatigue Condition
Behavioral: Control — time-matched task (sitting on the bike without pedalling)
  Arms: Control Condition

SUMMARY:
The main objective of this project is:

1. To assess the influence of physical fatigue on brain functioning during a balance and reaction time task in a healthy population. In a later stage, these experiments could be carried out in a clinical context (e.g. in an ankle sprain population).

The researchers will use a randomized, placebo controlled, counter-balanced, cross-over design. Twenty healthy subjects will visit the lab 3 times. On the first visit (familiarisation trial), the investigators will collect the participants' characteristics. The participants will also be familiarized to the procedures and materials of the experiment during this first visit. The second and third visit contain the experimental setup and will proceed as follows: first, the participants will fill in a pre-test checklist, a mental fatigue scale (M-VAS) and motivation scale. In the mean time a little blood will be collected from the ear lobe to determine lactate and glucose levels; also, blood pressure will be checked.

Next, the subjects will carry out a Y-balance test and a balance reaction-time test. Session rate of perceived exertion (SRPE) is measured to indicate how fatigued the participants feel due to the test battery; also, M-VAS is collected once more, as well blood lactate, glucose and blood pressure. These measures are followed by either a physical fatigue inducing task (Modified 30 seconds Wingate protocol) or time-matched control task (sitting on the bike without pedalling). Afterwards, researchers will collect blood lactate, glucose and blood pressure two times more; participants have to fill in M-VAS (2x), perform the same Y-balance test and balance reaction time test, and fill in the SRPE scale one more time. Heart frequency and EEG will be measured continuously during the trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological/cardiorespiratory/psychological/musculoskeletal disorders)
* Male and female
* No medication
* Non-smoker
* Between 18 and 35 years old

Exclusion Criteria:

* Back and/or lower extremity injuries during the past 6 months
* Bone/joint abnormalities
* Dizziness, history of loss of consciousness, any inner ear disorders
* Nervous system disorders or dysfunctions
* Uncorrected eye disorders/dysfunctions
* Illness
* Use of medication or any kind of drugs
* Use of alcohol, caffeine and heavy efforts 24 hours before each trial
* Not eating the same meal the night before and the morning of each experimental trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Y-balance test | Change in Y-balance performance: from baseline and 20 minutes after baseline (immediately after the assigned interventions)
  Balance and reach performance; participants have to maintain their balance while reaching as far as possible along 3 different directions
Balance-reaction time test | Change in balance and reaction time performance: from baseline and 20 minutes after baseline (immediately after the assigned interventions)
  Balance and reaction time performance; participants have to maintain their balance while reacting as fast as possible in 3 different directions.
EEG power spectrum analysis | Change in EEG power spectrum: from baseline and 20 minutes after baseline (immediately after the assigned interventions)
  Brain activity during the Y-balance test and balance-reaction time test will be registered at baseline and immediately after the assigned interventions.

SECONDARY OUTCOMES:
Mental fatigue Visual Analogue Scale (M-VAS) | Change in M-VAS: at baseline, 10 min after baseline (immediately after the first two balance tests), 15 min after baseline (immediately after the assigned interventions) and 25 min after baseline (immediately after the final 2 balance tests)
  Subjective measure of mental fatigue (0-10cm; 0 = no mental fatigue; 10 = maximal mental fatigue)
Perception of effort (Session RPE) | Change in session RPE: at baseline (immediately after the first two balance tests), and 15 min after baseline (immediately after the final 2 balance tests)
  Subjective measure of effort after completion of the test battery (scale from 0 to 10; 0 = very very easy; 10 = maximal effort)
Self-reported motivation | At baseline: prior to the first test battery
  Subjective measure of motivation assessed with the self-reported Motivation scale of Matthews et al.. (the questionnaire measures 2 constructs: intrinsic motivation and task succes motivation;the questionnaire comprises 14 questions scored from 0 to 4 [0 = not all motivated, while 4 = maximally motivated]. Each construct contains 7 questions).
Blood lactate | Blood lactate changes: at baseline, 10 min after baseline (immediately after the first two balance tests), 15 min after baseline (immediately after assigned interventions) and 25 min after baseline (immediately after the final two balance tests
  Capillary blood will be collected at the ear lobe for the determination of blood lactate (determined enzymatically)
Blood glucose | Blood glucose changes: at baseline, 10 min after baseline (immediately after the first two balance tests), 15 min after baseline (immediately after assigned interventions) and 25 min after baseline (immediately after the final two balance tests)
  Capillary blood will be collected at the ear lobe for the determination of blood glucose concentration
Blood pressure | Blood pressure change: at baseline, 10 min after baseline (immediately after the first two balance tests), 15 min after baseline (immediately after assigned interventions) and 25 min after baseline (immediately after the final two balance tests)
  Objective measure of blood pressure via eletronic blood pressure measuring device

CONTACTS AND LOCATIONS:
Overall Officials: Romain Meeusen, Professor, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No